CLINICAL TRIAL: NCT03886610
Title: Quantitative and Functional Longitudinal Multimodal Imaging of the Brain and Cervical Spinal Cord in Spinal Cord Injury: Correlation With Clinical Outcome
Brief Title: Association of Quantitative and Functional Imaging With Clinical Outcome After Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Collaborators: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Christiaanse Ernst, Radiologist, Swiss Paraplegic Research, Nottwil
Other Study IDs: 2018-37
Record Dates: First submitted 2019-03-21; First posted 2019-03-22 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy controls: Individuals without spinal cord injury
  Interventions: Other: Healthy controls
- Subacute SCI patients: Subacute patients with spinal cord injury (duration >2 weeks)
  Interventions: Other: Subacute SCI patients
- Chronic SCI patients: Patients with chronic spinal cord injury (duration ≥24 months)
  Interventions: Other: Chronic SCI patients

INTERVENTIONS:
Other: Healthy controls — individuals without spinal cord injury
  Groups: Healthy controls
Other: Subacute SCI patients — individuals with spinal cord injury ≥ 2 weeks
  Groups: Subacute SCI patients
Other: Chronic SCI patients — individuals with spinal cord injury ≥ 24 months
  Groups: Chronic SCI patients

SUMMARY:
The overall study aim is to provide additional magnetic resonance imaging parameters of the cervical spinal cord, brainstem and brain and a better understanding of changes after spinal cord injury (SCI) and to define new magnetic resonance (MR) biomarkers to correlate with sensomotoric functioning and clinical outcome.

DETAILED DESCRIPTION:
Injury of the spinal cord, for instance induced by trauma, is complex involving primary mechanisms caused by forces directly affecting the spinal cord and secondary mechanisms consisting of complex physiological processes after trauma.

Conventional magnetic resonance imaging (MRI) is the current standard to assess morphologic changes of the spinal cord after injury. However, conventional MRI provides little information regarding the health and integrity of the brain and spinal cord tissue itself, due to the fact that signal intensity changes are non-specific and do not correspond directly with physiological processes. This is reflected in the poor correlation of conventional MRI data with neurological and functional impairment in various spinal cord pathologies (such as multiple sclerosis compression myelopathy) and failure to provide reliable prognostic information.

By applying a combination of diffusion weighted imaging, functional MRI and magnetic resonance spectroscopy will give us a better understanding of the changes after injury of the cervical spinal cord, brainstem and brain. Correlating the imaging data with the neurological and clinical status of patients could improve the patient status prediction and therapy planning.

This study is divided into three sub-projects:

i) Reproducibility study of the MR measurements in healthy controls ii) Progression of MR biomarkers in subacute patients with SCI and comparison to chronic patients with SCI iii) Prediction of clinical outcome based on MR biomarkers

ELIGIBILITY:
Healthy controls:

Inclusion Criteria:

* age between 18 and 80 years
* no previous history of severe cervical trauma, traumatic brain injury, cervical surgery or signs of neurological impairment and no known neurological disease.

Exclusion Criteria:

* not meeting the MRI screening requirements
* unable to give consent
* unable to fulfill the above mentioned inclusion criteria

Subacute and chronic patients with spinal cord injury:

Inclusion Criteria:

* lesion level at or below C3
* etiology of the spinal cord injury is traumatic or non-traumatic
* age between 18 and 80 years
* time of trauma or onset of symptoms for subacute SCI patients is more than 3 weeks and for the chronic SCI patients more than 2 years

Exclusion Criteria:

* lesion level below L2
* other known pathology of the spinal cord/brain (e.g. MS) or progressive neurological disorders
* inability to meet the MRI screening requirements (e.g. pacemaker or other electronic devices),
* severe head trauma as defined by a Glasgow Coma Scale (GCS) of < 14
* patients who are ventilator dependant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * 20 healthy controls
  * 35 patients with subacute spinal cord injury
  * 20 patients with chronic spinal injury
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Fractional Anisotropy (FA) | 16-40 days after injury, 70-96 days after injury, 150- 186 days after injury
  Degree of anisotropy of a diffusion process (value between zero and one). A value of zero means that diffusion is isotropic, i.e. it is unrestricted (or equally restricted) in all directions. A value of one means that diffusion occurs only along one axis and is fully restricted along all other directions. FA is a measure often used in diffusion imaging where it is thought to reflect fiber density, axonal diameter, and myelination in white matter.

SECONDARY OUTCOMES:
Change in Apparent Diffusion Coefficient (ADC) | 16-40 days after injury, 70-96 days after injury, 150- 186 days after injury
  Measurement of the magnitude of diffusion (of water molecules) within tissue
Change in Relative Anisotropy (RA) | 16-40 days after injury, 70-96 days after injury, 150- 186 days after injury
  Measurement of the relative diffusion (of water molecules) within tissue

CONTACTS AND LOCATIONS:
Overall Officials: Ernst Christiaanse, MD, Principal Investigator — Swiss Paraplegic Centre
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Switzerland

IPD SHARING:
Plan to Share IPD: No